CLINICAL TRIAL: NCT05577819
Title: Prevalence and Prediction of Transthyretin Amyloidosis in Ambulatory Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Prevalence and Prediction of ATTR in Ambulatory Patients With HFpEF
Acronym: TTRinHFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Akcea Therapeutics (Industry); Pfizer (Industry); Alnylam Pharmaceuticals (Industry); Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Principal Investigator, Hanna Kim Gaggin, Principal Investigator, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P002061
Record Dates: First submitted 2021-07-16; First posted 2022-10-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Transthyretin Amyloidosis; Heart Failure; Heart Failure, Diastolic; Amyloidosis
Keywords: Transthyretin Amyloidosis; Heart Failure; Heart Failure, Diastolic; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Heart Failure; Heart Failure, Diastolic; Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients 65 and older with Heart Failure with Preserved Ejection Fraction (Experimental): Patients 65 years and older presenting to Massachusetts General Hospital with a known diagnosis of HFpEF and without a diagnosis of amyloidosis in the ambulatory (outpatient) setting will undergo a 99Tc-Pyrophosphate Scan to identify Cardiac Amyloidosis
  Interventions: Diagnostic Test: 99mTc-pyrophosphate Scintigraphy

INTERVENTIONS:
Diagnostic Test: 99mTc-pyrophosphate Scintigraphy — Cardiac Imaging Technique used to diagnose Transthyretin Cardiac Amyloidosis by use of 15 mCi of 99mTC-Pyrophosphate tracer
  Other Names: PYP Scan; Pyrophosphate Scan

SUMMARY:
Recent studies have shown that transthyretin amyloidosis (ATTR) can sometimes cause a type of heart failure where the pumping function of the heart is normal, also known as Heart Failure with Preserved Ejection Fraction (HFpEF) or diastolic heart failure. In this single center diagnostic study, we will evaluate for ATTR in patients with HFpEF in order to to determine how frequently this occurs and how we can predict which heart failure patients may have TTR amyloidosis. Our goal is to identify amyloidosis in heart failure patients earlier so that they can start treatment.

DETAILED DESCRIPTION:
Patients 65-years and older with HFpEF will be enrolled to participate in this single center, event driven (positive nuclear amyloid scan also known as 99mTc-pyrophosphate SPECT scan) study.

During the single study visit the following will be obtained:

* 99mTc-pyrophosphate SPECT scan
* Blood and DNA (optional) sample collection
* Questionnaires in regards to neuropathy, carpal tunnel, frailty, and Heart failure symptoms and how they may affect ones quality of life
* 6-Minute Walk Test
* ECG (electrocardiogram)
* Echocardiogram

Electronic health records will be reviewed for up to 5 years in order to determine hospitalization and survival of the study participants. Clinical outcomes of interest include a combined endpoint of days alive outside of the hospital from heart failure hospitalizations at one and five years, presence of autonomic neuropathy, presence of carpal tunnel syndrome, presence of polyneuropathy. Additionally, Individual clinical endpoints are also endpoints of interest.

The results from this study will be used to determine how frequently heart failure patients have transthyretin amyloidosis in their heart and better understand their symptoms. We hope that better understanding transthyretin amyloidosis in heart failure patients will help us identify affected patients so that they can receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of HFpEF.
* Age ≥65 years old

Exclusion Criteria:

* End stage chronic kidney disease on dialysis (CKD stage 5 as defined as eGFR <15mL/min)
* no history of HFrEF (LVEF<40%) with the exception of low LVEF in the setting of acute decompensation, AF RVR, ACS/MI, etc
* Negative 99mTc-pyrophosphate scan within a year
* Unable to lie down for 15 minutes for the 99mTc-pyrophosphate scan
* Known diagnosis of amyloidosis
* Severe valvular heart disease that is uncorrected (moderate to severe is considered exclusionary)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 515 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of 99mTc-pyrophosphate scan positive ATTR | Day 1 (day of study visit)
  A cardiac disease in which misfolded proteins aggregate into amyloid fibril and deposit interstitially, leading to diastolic dysfunction and heart failure

SECONDARY OUTCOMES:
New York Heart Association function classification | Day 1 (day of study visit)
  Classifies the severity of a patients Heart Failure in terms of their limitations during physical activity
Impact of HF as assessed by Kansas City Cardiomyopathy Questionnaire | Day 1 (day of study visit)
  Kansas City Cardiomyopathy Questionnaire is a questionnaire that determines in the impact of Heart Failure on their health status, such as quality of life, symptoms, function, etc.)
Exercise capacity as determined by a 6-minute walk test | Day 1 (day of study visit)
  The 6 minute walk test is used to determine an objective measurement of a patients aerobic capacity and endurance

OTHER OUTCOMES:
Presence of autonomic neuropathy | Time from study Visit until the date of documented event up to 5 years after the study closure
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events
Presence of carpal tunnel syndrome | Time from study Visit until the date of documented event up to 5 years after the study closure
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events
Presence of polyneuropathy | Time from study Visit until the date of documented event up to 5 years after the study closure
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events
Combined endpoint of days alive outside of hospital from HF hospitalizations at one and five years | Time from study Visit until the date of documented event up to 5 years after the study closure
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events
Individual endpoints of all-cause mortality, cardiovascular mortality, all-cause hospitalizations, cardiovascular hospitalizations and HF hospitalizations. | Time from study Visit until the date of documented event up to 5 years after the study closure
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events

CONTACTS AND LOCATIONS:
Overall Officials: Hanna K Gaggin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided